CLINICAL TRIAL: NCT05463302
Title: Investigating the Efficacy of Sleepgift Blanket on Sleep Quality and Heart Health
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: BB Holistics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Sleep Gift Blanket
Record Dates: First submitted 2022-07-12; First posted 2022-07-18 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2023-12

CONDITIONS: Sleep
Keywords: electromagnetic field effect; sleep quality; EMF blocker
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: it is two period design with one cross over
Who Masked: Participant
Masking Description: participants receive two similar blankets, while one of them is real and one is sham but they are blind to which one is which.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active EMF blanket (Active Comparator): participants will receive the real EMF blocker blanket
  Interventions: Device: Active sleepgift blanket; Device: Sham Sleepgift Blanket
- Sham EMF blanket (Placebo Comparator): participants will receive the sham EMF blocker blanket
  Interventions: Device: Active sleepgift blanket; Device: Sham Sleepgift Blanket

INTERVENTIONS:
Device: Active sleepgift blanket — Participants for group1 will be provided with real/active sleepgift blanket first for 10 consecutive nights and then cross over.
Device: Sham Sleepgift Blanket — Participants for group 2 will be provided with sham sleepgift blanket for 10 consecutive nights and then cross over.

SUMMARY:
Exposure to electromagnetic field (EMF) emitted by mobile phones and devices with WIFI is on the rise and so is the EMF effects on sleep quality and well-being of individuals with high exposures to EMF. Some studies have shown poor sleep quality among individuals with long-term occupational exposure to EMF, and some have shown association between EMF long-term exposure and neuropsychiatric disorders including depression. This study aims to investigate a commercially available EMF- blocker blanket, called Sleepgift, that claims helping people to have a better sleep and improved health. We will investigate the Sleepgift efficacy on adults' quality of sleep and their vital signals as a measure of their well-being in a placebo-controlled single- blind cross-over designed study. Participants will sleep in our sleep lab at baseline and then 10 days later with the Sleepgift blanket after using it every night for the past 10 consecutive days. Participants will be given two blankets for each cycle of the study as it is a cross-over designed study: one Sleepgift and one regular blanket; they will not know which one is real or sham. There will be one-month washout period between the two cycles of the cross-over study. We aim to enroll 30 adults for the study. Participants' sleep quality will be measured by the established device called Prodogy; their vital signals will also be measured and monitored through the night. The collected data will be analyzed statistically for any significant effect of the Sleepgift blanket on sleep quality and vital signals such as heart's rhythm and heart rate variability.

ELIGIBILITY:
Inclusion Criteria:

* 18 y<age<70 years
* Being generally healthy (cognitively and psychologically)
* ability to read, write and speak English fluently.

Exclusion Criteria:

* Being diagnosed with any neurological, intellectual disability, major depression/anxiety, bipolar disorder, schizophrenia or any other major mood disorder.
* Inability to adequately communicate in English
* Current substance abuse disorder
* Currently participating in another therapeutic study
* Being on a regular pain killer, sleeping or depression pill.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2024-10-11 (Actual)

PRIMARY OUTCOMES:
Sleep quality measure | Through study completion, 2 years approximately
  The change in the value of Odds of the Product (ORP) from baseline line to post-intervention, measured by the Prodigy device which is a combination of the EEG band waves. ORP is only one value output of the device.

SECONDARY OUTCOMES:
heart rate variability | Through study completion, 2 years approximately
  the change in heart rate variability (HRV) measured from beat to beat R-R interval.

CONTACTS AND LOCATIONS:
Overall Officials: Zahra Moussavi, Ph.D., Principal Investigator — University of Manitoba
Locations (1):
- Riverview Health Center, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Yes
When the study is finished, de-identified data could be shared publicly by other researchers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After Aug. 2025